CLINICAL TRIAL: NCT07161388
Title: Durvalumab Consolidation After Chemoradiation Therapy (CRT) for Patients With Limited Stage Small-Cell Lung Cancer in China: A Multicentre, Observational Study (DREAM)
Brief Title: Durvalumab Consolidation After Chemoradiation Therapy for Limited Stage SCLC in China
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419QR00019
Record Dates: First submitted 2025-09-05; First posted 2025-09-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Limited Stage Small-Cell Lung Cancer
Keywords: SCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LS-SCLC: Patients with LS-SCLC who received platinum-based cCRT/sCRT followed by durvalumab consolidation as first line treatment at the discretion of physicians.

SUMMARY:
This prospective, multicentre, observational study aims to assess the effectiveness and safety of durvalumab as consolidation treatment for patients with LS-SCLC who have not progressed following CRT in real-world setting.

DETAILED DESCRIPTION:
In this study, the effectiveness and safety profile of durvalumab consolidation following CRT in patients with LS-SCLC will be investigated in a real-world setting. Clinical outcomes will be explored across different CRT modalities and regimens according to local practice. Additionally, evidence will be generated on durvalumab consolidation following CRT regardless of concurrent or sequential setting. The subsequent treatment patterns of patients who experience disease progression during or after durvalumab consolidation will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Age ≥18 years
* Histologically or cytologically documented LS-SCLC (Stage I-III SCLC [T any, N any, M0] according to the American Joint Committee on Cancer Staging Manual [AJCC Cancer Staging Manual, 8th Edition], that can be safely treated with definitive radiation doses. Excludes T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan)
* ECOG PS 0-2 (prior to the first dose of durvalumab after CRT)
* No disease progression following cCRT/sCRT (cCRT refers to chemotherapy and radiotherapy are administered with overlap; sCRT refers to chemotherapy and radiotherapy are delivered in a sequential manner with no overlap)
* Patients who received platinum-based cCRT/sCRT followed by durvalumab consolidation as first-line treatment at the discretion of physicians are eligible (the time interval from the end of cCRT/sCRT to the first dose of durvalumab consolidation should be within 3 months)

  * Patients who started durvalumab consolidation ≤3 months before enrolment in the study will be allowed (irrespective of whether they continue to receive durvalumab at time of enrolment or already discontinued treatment)

Exclusion Criteria:

* Patients treated with CRT only without subsequent durvalumab consolidation
* Patients received durvalumab or any other anti-PD-1/anti-PD-L1 antibodies along with CRT
* Patients who previously were involved, or currently are, or plan to be involved in any other interventional anti-cancer clinical studies for LS-SCLC
* Prior exposure to immune-mediated therapy including, but not limited to, other anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines
* Judgment by the investigator that the patient should not participate in the study because the patient is unlikely to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients (with age ≥18 years old) who able to provide informed consent received platinum-based cCRT/sCRT followed by durvalumab consolidation as first-line treatment at the discretion of physicians and no disease progression following cCRT/sCRT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
rwPFS | From 3 months before enrolment to follow-up of up to 36 months
  From date of first dose of durvalumab consolidation treatment until progression as assessed in real-world, or death due to any cause.
  The primary measure of interest is the median rwPFS.

SECONDARY OUTCOMES:
TTD | From 3 months before enrolment to follow-up of up to 36 months
  From date of first dose of durvalumab consolidation treatment until discontinuation of treatment for any reason, including disease progression, toxicity and death.
  The measure of interest is the median TTD.
OS | From 3 months before enrolment to follow-up of up to 36 months
  From first dose of durvalumab consolidation treatment until the date of death due to any cause. 6, 12, 18, and 24-months landmark rate of OS will be described.

OTHER OUTCOMES:
TRAE, SAE, irAE, other AEs | From 3 months before enrolment to follow-up of up to 36 months
  Treatment-related adverse event (TRAE), serious adverse event (SAE), immune-related adverse events (irAE), adverse events (AEs) leading to durvalumab dose interruption, discontinuation and AEs leading to death.
TFST | From 3 months before enrolment to follow-up of up to 36 months
  From date of first dose of durvalumab consolidation treatment until the start date of the first subsequent anti-cancer therapy after discontinuation of durvalumab, or death due to any cause. Median TFST will be described.
Patterns of progression and post-progression therapy. | From 2 months before enrolment to follow-up of up to 35 months
  Number and percentage of subjects with certain progression sites will be described.
rwPFS in subgroups | From 3 months before enrolment to follow-up of up to 36 months
  rwPFS will be analysed within pre-specified subgroups.
Baseline characteristics | During enrolment period up to 12 months
  To describe baseline characteristics of patients who received prior cCRT and sCRT including the time from diagnosis to starting durvalumab and the time from the end of radiation to starting durvalumab.

CONTACTS AND LOCATIONS:
Overall Officials: JinMing Yu, Doctor, Principal Investigator — Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital)
Locations (21):
- China (21):
  - Research Site, Beijing
  - Research Site, Cangzhou
  - Research Site, Dongguan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Huzhou
  - Research Site, Jinan
  - Research Site, Jinzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Tianjing
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Yangzhou
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/